CLINICAL TRIAL: NCT05101993
Title: Long-term Follow-up on LAA Exclusion Using AtriClip, VCLIP Post-Market Study, CLINICAL TRIAL PROTOCOL: CP-2021-03
Brief Title: VCLIP Post-Market Study, Long-term Follow-up on LAA Exclusion Using AtriClip
Acronym: VCLIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-2021-03
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2023-04

CONDITIONS: Left Atrial Appendage Absent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- AtriClip group (Experimental): Subjects eligible for evaluation are those who had undergone designated non-emergent, cardiac surgical procedure(s), received an AtriClip implant (with devices under investigation) and who were willing to return for follow-up chest imaging to ascertain Left Atrial Appendage (LAA) exclusion and met inclusion exclusion criteria.
  Interventions: Device: AtriClip

INTERVENTIONS:
Device: AtriClip — Received AtriClip for exclusion of left atrial appendage during concomitant cardiac procedure

SUMMARY:
Retrospective-prospective, multi-center, non-randomized, unblinded, post-market study to evaluate the long-term performance and safety of AtriClip® FLEX-V LAA and PRO•V LAA Exclusion devices for exclusion of the left atrial appendage of the heart during concomitant cardiac procedures.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the long-term performance and safety of AtriClip® FLEX-V LAA and PRO•V LAA Exclusion devices for exclusion of the left atrial appendage of the heart during concomitant cardiac procedures in participants for which a VCLIP was placed previously. Participants are consented and evaluated to confirm long-term performance of the AtriClip®.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is greater than or equal to 18 years of age.
2. Subject who received the AtriClip FLEX-V or PRO•V implant during a non-emergent cardiac surgical procedure
3. Subject is willing and able to provide written informed consent
4. Subject is willing and able to return for scheduled follow-up visit and imaging (CTA or TEE)

Exclusion Criteria:

1. Inability, unwillingness, or contraindication to undergo TEE or CTA imaging
2. Subjects who are pregnant or breast feeding
3. Subjects with active COVID-19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Zias, MD, Principal Investigator — NYU Langone Health
Locations (11):
- United States (11):
  - Franciscan Health, Indianapolis, Indiana
  - Washington University School of Medicine, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - NYU, New York, New York
  - Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - Mercy Health Cincinnati, Cincinnati, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Prisma Health, Greenville, South Carolina
  - Centra Lynchburg General Hospital, Lynchburg, Virginia
  - Aurora Research Institute LLC, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AtriClip Group
Started | 156
Completed | 155
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Participants Enrolled
Arm/Group | AtriClip Group
Number analyzed (Participants) | 155
Age, Categorical [Count of Participants; unit: Participants] — Population: 1 subject withdrew participation prior to index procedure
  Participants
    <=18 years | 0
    Between 18 and 65 years | 61
    >=65 years | 94
Age, Continuous [Median (Full Range); unit: years] — Population: 1 subject withdrew participation before index procedure
  years | 66 [41 to 85]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: 1 subject withdrew participation prior to index procedure
  Participants
    Female | 34
    Male | 121
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 1 subject withdrew participation before index procedure
  Participants
    White | 146
    Black | 5
    Asian | 2
    Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Primary Performance Endpoint
Description: Left Atrial Appendage exclusion defined as absence of residual communication (≤3 mm residual communication with LAA) between the left atrium (LA) and the LAA as assessed by CTA or TEE imaging at the last follow-up visit. The images will be reviewed by an independent core lab using a standardized imaging protocol.
Time Frame: 12-months or greater post-procedure, an average of 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | AtriClip Group
Number analyzed (Participants) | 151
Participants | 151

2. Primary Outcome: Primary Safety Endpoint
Description: Incidence of the following serious adverse events within 30-days, if related tot he device and/or implant procedure:
  * Death
  * Ischemic Stroke
  * Transient Ischemic Attack
  * Systemic Embolism
  * Hemorrhagic Stroke
  * Major Bleeding (BARC 3 and above)
  * Surgical site infection
  * Pericardial effusion requiring intervention
  * Clinical diagnosis of myocardial infarction
Time Frame: 30-days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | AtriClip Group
Number analyzed (Participants) | 155
Participants | 0
Statistical Analysis 1: Comparison: AtriClip Group; Test type: Superiority; p < 0.0001, Chi-squared

3. Secondary Outcome: Performance
Description: A residual LAA neck ≤10 mm as assessed by CTA or TEE imaging at the last follow-up visit
Time Frame: 12-months or greater post-procedure, an average of 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | AtriClip Group
Number analyzed (Participants) | 152
Participants | 135

4. Secondary Outcome: Long-term Thromboembolic Events
Description: Incidence of thromboembolic events (ischemic stroke, TIA, systemic embolism) of any cause through the last follow-up visit.
Time Frame: 12-months or greater post-procedure, an average of 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | AtriClip Group
Number analyzed (Participants) | 155
Participants | 0

5. Secondary Outcome: Device and Procedure Long-term Safety
Description: Number of Participants with Device or Procedure Related SAEs through the last follow-up visit
Time Frame: 12-months or greater post-procedure, an average of 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | AtriClip Group
Number analyzed (Participants) | 155
Participants | 5

ADVERSE EVENTS:
Time Frame: 12-months or greater post-procedure, an average of 1.5 years
Description: Serious Adverse Events
Arm/Group | AtriClip Group
All-Cause Mortality (participants affected / at risk) | 0/155
Serious Adverse Events (participants affected / at risk) | 76/155
Other Adverse Events (participants affected / at risk) | 0/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AtriClip Group (N=155)
Arrhythmia Needing Medical Treatment (new onset) (Cardiac disorders) | 9
Pleural Effusion (Blood and lymphatic system disorders) | 7
Bleeding Event (Blood and lymphatic system disorders) | 3
GI Bleed (Gastrointestinal disorders) | 3
Hernia (Musculoskeletal and connective tissue disorders) | 4
Sepsis (Immune system disorders) | 3
Angina (Cardiac disorders) | 2
Bowel Obstruction (Gastrointestinal disorders) | 3
Vascular Disease (Cardiac disorders) | 3
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Conduction Disturbance (Immune system disorders) | 2
Congestive Heart Failure (Cardiac disorders) | 2
Myocardial Infraction (Cardiac disorders) | 2
Pericardial Effusion (Cardiac disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
TIA or Neurological Deficit (Nervous system disorders) | 2 — (lasting <24h) without Infraction
Aphasia (Nervous system disorders) | 1
Atrial Fibrillation with Rapid Ventricular rate (Cardiac disorders) | 1
AV block requiring permanent pacemaker (new onset) (Cardiac disorders) | 1
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Infection (Infections and infestations) | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1
Left foot partial 1st ray amputation (Surgical and medical procedures) | 1
Nausea and Abdominal Pain-Dehydration (General disorders) | 1
Pericarditis (Cardiac disorders) | 1
Post operative ileus requiring decompressive colonoscopy (Surgical and medical procedures) | 1
Pulmonary Embolism (Cardiac disorders) | 1
Renal Insufficiency (Renal and urinary disorders) | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Sinus Node Dysfunction (Cardiac disorders) | 1
Sternal Dehiscence (Cardiac disorders) | 1
Stroke, Other (Cardioembolic) (Cardiac disorders) | 1
Stroke, Ischemic (Cardiac disorders) | 1
Thrombus (Cardiac disorders) | 1
Thrombocytopenia (Cardiac disorders) | 1
Tricuspid Valve Regurgitation (Cardiac disorders) | 1
Excessive Bleeding r/t Procedure (req >2u Blood or intervention) (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT05101993/Prot_SAP_000.pdf